CLINICAL TRIAL: NCT02673476
Title: A Phase 2a, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Orally Administered ALS-008176 in Adults Hospitalized With a Respiratory Syncytial Virus-Related Illness
Brief Title: A Phase 2a Study to Evaluate Orally Administered ALS-008176 in Adults Hospitalized With a Respiratory Syncytial Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALS-8176-510
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Identical Placebo Comparator
  Interventions: Drug: Placebo
- ALS-008176 (Experimental): ALS-008176 tablets
  Interventions: Drug: ALS-008176

INTERVENTIONS:
Drug: ALS-008176 — ALS-008176 tablets
  Arms: ALS-008176
Drug: Placebo — Identical placebo tablets
  Arms: Placebo

SUMMARY:
This study is being to see how effective and safe ALS-008176 is in treating adults in the hospital with a Respiratory Syncytial Virus-Related Illness.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥50 years of age.
2. Female subjects of non-childbearing potential (i.e., surgically sterilized, post-menopausal [amenorrhea for 1 year confirmed by negative hormone panel]) who also have a negative pregnancy test at screening.
3. Male subjects must be either surgically sterilized (e.g., post-vasectomy or orchiectomy) or willing to adhere to the study's contraceptive requirements. Male subjects'female partner(s) must be surgically sterilized or post-menopausal (amenorrhea for 1 year) or their female partner(s) of child-bearing potential must be willing and able to adhere to the contraceptive requirements.
4. Each subject or their legal guardian must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study before starting any screening activities.
5. Subject has a positive RT-PCR test result for RSV at the time of screening. NOTE: Co-infection with other acute viruses or bacteria is permitted.
6. Subject has been, or will be, admitted to the hospital for an acute respiratory illness with signs and symptoms consistent with a viral infection (e.g., fever, cough, nasal congestion, runny nose, sore throat, myalgia, lethargy, shortness of breath, or wheezing) with onset <7 days from the anticipated time of randomization.

Exclusion Criteria:

1. Subject is undergoing peritoneal dialysis, hemodialysis or hemofiltration or has an estimated glomerular filtration rate (GFR, determined by Cockcroft-Gault Formula) <30 mL/min.
2. Subject has presence of any concurrent illness, including laboratory, vital sign, ECG, or physical exam findings, or medical history that, in the opinion of the investigator, would place the subject at an unreasonably increased risk as a result of participation in this study.
3. Subject reports receiving an investigational drug or vaccine within 30 days, or 5 half-lives (whichever is longer) prior to the planned first dose of study drug.
4. Subject has a known history of human immunodeficiency virus (HIV) or chronic, active hepatitis infection.
5. ALT >3×ULN AND bilirubin >2×ULN (direct >35%) OR ALT>5×ULN
6. Subjects who have been hospitalized for >72 hours at the time of randomization.
7. Subjects anticipated to be hospitalized for <24 hours after randomization.
8. Subjects who are not expected to survive for <48 hours.
9. Recent (<5 half-lives) use, or anticipated use during conduct of the study, of concomitant medications (prescription and non-prescription) which are inhibitors of the OAT3 transporter.
10. Treatment of the current illness with drugs specifically targeting the RSV infection itself (e.g., RSV immunoglobulin, ribavirin, palivizumab). Medications treating the sequelae of the RSV infection or any concurrent illness are permitted if not otherwise excluded.
11. Subjects unwilling to undergo regular nasal swab procedures or with any physical abnormality which limits the ability to collect regular nasal specimens.
12. Subjects that are considered by the investigator to be immunocompromised over the past 12 months, whether due to underlying medical condition or medical therapy.
13. Subjects unable to take medications enterally (e.g., orally or via nasogastric or PEG tube) or a known gastrointestinal-related condition that may interfere with study drug absorption.
14. Female subject that is pregnant or breastfeeding
15. In the investigator's opinion, the subject is unwilling or unable to comply with protocol requirements, instructions, and protocol stated restrictions, and is unlikely to complete the study as planned.
16. Subject has known or suspected hypersensitivity to the study drug or its excipients (microcrystalline cellulose, mannitol, croscarmellose sodium, magnesium stearate, polyethylene glycol, polyvinyl alcohol, talc, titanium dioxide).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
AUC of RSV RNA | From prior to first dose to study day 7
  Area under the curve (AUC) of RSV ribonucleic acid (RNA) from nasal swabs immediately prior to 1st dose of study drug (baseline) until Day 7.

SECONDARY OUTCOMES:
Time from baseline to non-detectability of RSV from nasal swab | From prior first dose to study day 28
  Time from baseline to non-detectability of RSV from nasal swab
Percent of subjects with undetectable RSV by qPCR | From study day 3, and every two days until study day 7
  Percent of subjects with undetectable RSV by qPCR on Day 3, Day 5, and every other day until 2 days after last dose from nasal swab
Peak post-baseline viral load | From before first dose to study day 28
  Peak post-baseline viral load from nasal swab
Rate of decline from baseline in viral load during treatment from nasal swab | From before first dose to study day 2
  Rate of decline from baseline in viral load during treatment from nasal swab
Duration of hospital stay | From first dose to study day 28
  Duration of hospital stay
Safety data: Composite number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG, echo and abnormal clinical laboratory results | From screening to study day 28
  Tabulation of the number and frequency of treatment emergent adverse events, physical examination findings, abnormal vital signs, 12 lead ECG, echo and abnormal clinical laboratory results (including chemistry, hematology, and urine).
PK parameters: Cmax | From first dose to study day 28
  PK parameters in plasma following repeat dose administration: Cmax
PK parameters: tmax | From first dose to study day 28
  PK parameters in plasma following repeat dose administration: tmax
PK parameters: AUClast | From first dose to study day 28
  PK parameters in plasma following repeat dose administration: AUClast
PK parameters: t1/2 | From first dose to study day 28
  PK parameters in plasma following repeat dose administration: t1/2
PK parameters: AUC0 tau | From first dose to study day 28
  PK parameters in plasma following repeat dose administration: AUC0 tau

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Oey, Study Director — Alios Biopharma Inc.
Locations (21):
- United States (11):
  - Lake Internal Med. Assoc., Eustis, Florida
  - The Research Center, Inc., Hialeah, Florida
  - JDH Medical Group LLC, Miami, Florida
  - St Lucie Medical Center, Port Saint Lucie, Florida
  - Tampa Genereal Hospital, Tampa, Florida
  - Infectious Disease Specialists of Atlanta, Atlanta, Georgia
  - Kentucky Lung Clinic, PSC, Hazard, Kentucky
  - Bronson Methodist Hosp. Ped, Kalamazoo, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - University of Missouri- Clinical Research Center, Columbia, Missouri
  - Washington Univ School of Med, St Louis, Missouri
- Australia (7):
  - Westmead Hospital, Northmead, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Heal.-Monash Lung&Sleep, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Wellington Regional Hospital, Newtown, Wellington Region, New Zealand
- Raffles Hospital, Singapore, Singapore
- Taipei Med. Uni-Shuang Ho Hosp, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No data will be shared